CLINICAL TRIAL: NCT03696043
Title: Application of Image Guidance Technology to Bedside External Ventricular Drain Placement
Brief Title: External Ventricular Drain Placement Stealth Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1487; A535700 (Other: UW Madison); SMPH/NEURO SURG/NEURO SURG (Other: UW Madison); Protocol Version 8/8/2024 (Other: UW Madison)
Record Dates: First submitted 2018-05-24; First posted 2018-10-04 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: External Ventricular Drain; Intracranial Pressure
Keywords: intracranial pressure; external ventricular drain; cerebrospinal fluid

STUDY DESIGN:
Intervention Model Description: Target of 100 participants - 50% freehand EVD placement and 50% image guided EVD placement. Randomization is every other patient will received image guided EVD placement
Who Masked: Participant
Masking Description: Target of 100 participants - 50% freehand EVD placement and 50% image guided EVD placement. Randomization is every other patient will received image guided EVD placement
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVD placement (Active Comparator): Catheter placement is most commonly performed via a freehand approach using external anatomical landmarks to help identify the location of the lateral ventricle within the brain without the aid of imaging. Proper identification of the ventricles on pre-procedure imaging, surgeon skill, and estimation of pathologic perturbations to the normal location of the ventricles all factor into the success of catheter placement. Multiple passes are often required. The accuracy rate from the freehand technique has been reported to range from 40 to 98 percent.
  Interventions: Other: EVD placement
- Axium Stealth Image Guidance (Experimental): The novelty of this study is to investigate whether using image guidance technology can improve EVD catheter placement. Image guidance is used very commonly for EVD and shunt placement in the operating room with excellent accuracy and precision. We hypothesize that using this same workflow at the bedside will improve accuracy; decrease the number of passes needed for a successful placement, decrease the number of post-placement hemorrhagic events, and help improve the effectiveness of the catheter as well as patient outcomes.
  Interventions: Other: Axium Steatlh Image Guidance; Other: EVD placement

INTERVENTIONS:
Other: Axium Steatlh Image Guidance — The Axiem Stealth imaging guidance system uses a probe (AxiEM Registration Probe) and a side mount emitter (AxiEM Side Mount Emitter) to register the patient's head in relation to the probe. A trajectory (entry point and target) is then planned. This registration process takes an estimated 5-15 minutes to perform. A separate stylet (StealthStation EM Stylet) is designed specifically for the catheter and slides down the center of the catheter. A burr-hole is created at the predefined precise location and the catheter is passed to the target under electromagnetic guidance.
  Arms: Axium Stealth Image Guidance
Other: EVD placement — A sterile field is prepared about 10-12 centimeters posterior to the eye and about 2-3 cm lateral to the midline of the skull. An incision is made at this point and a burr hole is created using a hand drill. The catheter is advanced in a trajectory perpendicular to the skull, which results in a direction that is towards the ipsilateral medial canthus and ipsilateral tragus which are other landmarks that can be used.

SUMMARY:
External ventricular drain (EVD) placement is performed very often in neurosurgical practices. EVD's are most commonly placed at the bedside using external anatomical landmarks to guide the catheter into the frontal horn of the ipsilateral lateral ventricle. EVDs are often placed due to acute neurological compromise and require timely insertion.

Accurate catheter placement is essential to achieving effective external CSF drainage without complications or occlusion/failure of the catheter. Catheter placement is most commonly performed via a freehand approach using external anatomical landmarks to help identify the location of the lateral ventricle within the brain without the aid of imaging. Proper identification of the ventricles on pre-procedure imaging, surgeon skill, and estimation of pathologic perturbations to the normal location of the ventricles all factor into the success of catheter placement. Multiple passes are often required. The accuracy rate from the freehand technique has been reported to range from 40 to 98 percent.

Current methods for EVD placement do not compensate for superficial brain vessels or pathology that may alter the intracranial anatomy such as trauma, hemorrhage, or mass lesions. Some studies have attempted to use CTA imaging to identify intracranial vessels in an attempt to avoid them during placement.

Image guidance is a tool used very commonly for placement of EVD's and shunts in the operating room. AxiEM Stealth is a noninvasive image localization modality that registers a CT or MRI to the individual patients facial and scalp anatomy.

This study will compare the current standard of care of freehand placement of bedside external ventricular catheters to the placement of EVD catheters with AxiEM Stealth image guidance.

DETAILED DESCRIPTION:
External ventricular drain (EVD) placement is performed very often in neurosurgical practices. EVD's are used most commonly to monitor intracranial pressure and divert cerebrospinal fluid (CSF) in patients with increased intracranial pressures. Pathologies where EVDs are most frequently needed include hydrocephalus, malignancy, and/or trauma. EVD's are most commonly placed at the bedside using external anatomical landmarks to guide the catheter into the frontal horn of the ipsilateral lateral ventricle. EVDs are often placed due to acute neurological compromise and require timely insertion. This can increase the associated risk and result in complications.

Accurate catheter placement is essential to achieving effective external CSF drainage without complications or occlusion/failure of the catheter. Catheter placement is most commonly performed via a freehand approach using external anatomical landmarks to help identify the location of the lateral ventricle within the brain without the aid of imaging. Proper identification of the ventricles on pre-procedure imaging, surgeon skill, and estimation of pathologic perturbations to the normal location of the ventricles all factor into the success of catheter placement. Multiple passes are often required. The accuracy rate from the freehand technique has been reported to range from 40 to 98 percent. A very basic grading scale has been developed to assess placement but does not include items such as the number of passes until successful placement and presence of post placement hemorrhage or other neurological complications. An increased number of passes increases the risk of post placement hemorrhage and may damage the brain. Hemorrhage has been reported to occur after catheter placement at rates ranging from 0.2 to 41 percent.

Current methods for EVD placement do not compensate for superficial brain vessels or pathology that may alter the intracranial anatomy such as trauma, hemorrhage, or mass lesions. Some studies have attempted to use CTA imaging to identify intracranial vessels in an attempt to avoid them during placement.

Image guidance is a tool used very commonly for placement of EVD's and shunts in the operating room. AxiEM Stealth is a noninvasive image localization modality that registers a CT or MRI to the individual patients facial and scalp anatomy. A probe can then be used to identify, in real-time, the underlying anatomy and trajectories. This imaging guidance may improve the accuracy of EVD placement.

This study will compare the current standard of care of freehand placement of bedside external ventricular catheters to the placement of EVD catheters with AxiEM Stealth image guidance. Accuracy of the tip of the catheter, occurrence of post-placement hemorrhage, the number of passes required for CSF flow, ventricle diameter, catheter clogging/failure, time required for placement, patient demographics and other secondary outcome measures such as Glasgow Outcome Scale (GOS) and Modified Rankin Score (MRS) will be collected. The hypothesis is that image guided EVD catheter placement will improve accuracy, decrease the number of brain transgressions, and decrease complications of EVD placement.

What makes up an external ventricular drain and how does it work? An external ventricular drain (EVD) is comprised of a catheter, drainage tubing, and a collection system. Once the catheter is in the ventricular system, it works by measuring the intracranial pressure via a transducer and drains excess CSF from the ventricular system to ensure pressures does not exceed a set threshold. Normal intracranial pressures range from about 5-20 mmHg and are usually around 10mmHg. The EVD system can be set at a certain level and when the intracranial pressures rise above that level, CSF drains out the catheter into the collecting system. The EVD system can be raised or lowered to create different intracranial pressure thresholds and keep intracranial pressures controlled in patients that have a pathology, such as cerebral swelling or ventricular obstruction, leading to increased pressures.

What is the current technique used to place an EVD? A sterile field is prepared about 10-12 centimeters posterior to the eye (either right or left as clinically indicated) and about 2-3 cm lateral to the midline of the skull. This point should be about 1 cm anterior to the coronal suture. An incision is made at this point and a burr hole is created using a hand drill. The EVD catheter is prepared using a stylet to help with movement through the brain parenchyma. The catheter is advanced in a trajectory perpendicular to the skull, which results in a direction that is towards the ipsilateral medial canthus and ipsilateral tragus which are other landmarks that can be used. The catheter is advanced to 5-6 cm and the stylet is removed to assess for CSF flow. If CSF flow is not appreciated, then the catheter is passed softly for about 1 more centimeter. If CSF flow is still not appreciated, the catheter is removed and the stylet replaced for another attempt. If unsuccessful after 3 attempts, the catheter can be left in place and a head CT can be done to assess the adjustments that need to be made. This can often take up to 10 passes or more if there is significant brain shift due to mass effect or aberrant anatomy. Once CSF flow is obtained, the catheter is tunneled posteriorly and anchored to the skin with a stitch. The incision is then closed and the catheter is connected to the drainage tubing of the collection system. The presence of CSF drainage is checked at multiple points during closure to ensure that the catheter remains in good position.

How does Axiem Stealth work as an image guidance system and how is it used for EVD placement? The first step for using the image guidance system is to upload the most recent (since admission or within 6 hours from bleeding) head CT or MRI into the Stealth station that has been obtained since admission. The Axiem Stealth imaging guidance system uses a probe (AxiEM Registration Probe) and a side mount emitter (AxiEM Side Mount Emitter) to register the patient's head in relation to the probe. A trajectory (entry point and target) is then planned. This registration process takes an estimated 5-15 minutes to perform. A separate stylet (StealthStation EM Stylet) is designed specifically for the catheter and slides down the center of the catheter. A burr-hole is created at the predefined precise location and the catheter is passed to the target under electromagnetic guidance.

Relevance of this research:

The novelty of this study is to investigate whether using image guidance technology can improve EVD catheter placement. Image guidance is used very commonly for EVD and shunt placement in the operating room with excellent accuracy and precision. The hypothesis is that using this same workflow at the bedside will improve accuracy; decrease the number of passes needed for a successful placement, decrease the number of post-placement hemorrhagic events, and help improve the effectiveness of the catheter as well as patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bedside external ventricular drain placement determined by attending physician
* Age ≥ 18 years and ≤ 88 years
* Male or Female
* Patients or consentable family member must sign a written informed consent prior to EVD placement
* Stealth compatible head CT or MRI

Exclusion Criteria:

* Patients ≤ 18 and ≥ 88 years of age
* Prisoner status
* Subjects who decline participation into the study
* Subjects determined to be medically or neurologically to high of a risk for the study, determined by attending physician
* Patients who undergo emergent EVD placement via emergency consent
* Subjects for whom self-consent or consent by a LAR cannot be obtained or cannot be obtained
* Pregnant women
* Non-English speaking patients

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of catheter passes or attempts | baseline
  Collection of number of passes needed for successful catheter placement
Accuracy of catheter tip compared to foramen of Monro | baseline
  Measurement of accuracy for catheter tip compared to foramen of Monro with accuracy formula

SECONDARY OUTCOMES:
Occurrence of post-placement hemorrhage | baseline and 12 months
  Anotation of occurrence of hemorrhage post-catheter placement by either freehand or image guided
New neurological deficits | baseline and 12 months
  Utilization of the Glasgow Come Score and mRS scale to measure new neurological symptoms
Durability of EVD | baseline and 12 months
  Presence of clogging/ failure
Time required catheter insertion | baseline
  Anotation of time allocation for catheter insertion - both methods
Infection rate | baseline and 12 months
  Occurrence of ventriculostomy infection (meningitis, ventriculitis, cerebritis)

CONTACTS AND LOCATIONS:
Overall Officials: Azam Ahmed, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patil V, Lacson R, Vosburgh KG, Wong JM, Prevedello L, Andriole K, Mukundan S, Popp AJ, Khorasani R. Factors associated with external ventricular drain placement accuracy: data from an electronic health record repository. Acta Neurochir (Wien). 2013 Sep;155(9):1773-9. doi: 10.1007/s00701-013-1769-y. Epub 2013 May 23. PMID 23700258
- [Background] Mahan M, Spetzler RF, Nakaji P. Electromagnetic stereotactic navigation for external ventricular drain placement in the intensive care unit. J Clin Neurosci. 2013 Dec;20(12):1718-22. doi: 10.1016/j.jocn.2013.03.005. Epub 2013 Aug 30. PMID 23993898
- [Background] Patil V, Gupta R, San Jose Estepar R, Lacson R, Cheung A, Wong JM, Popp AJ, Golby A, Ogilvy C, Vosburgh KG. Smart stylet: the development and use of a bedside external ventricular drain image-guidance system. Stereotact Funct Neurosurg. 2015;93(1):50-8. doi: 10.1159/000368906. Epub 2015 Jan 31. PMID 25662506
- [Background] Sarrafzadeh A, Smoll N, Schaller K. Guided (VENTRI-GUIDE) versus freehand ventriculostomy: study protocol for a randomized controlled trial. Trials. 2014 Dec 5;15:478. doi: 10.1186/1745-6215-15-478. PMID 25480528
- [Background] Robertson FC, Abd-El-Barr MM, Mukundan S Jr, Gormley WB. Ventriculostomy-associated hemorrhage: a risk assessment by radiographic simulation. J Neurosurg. 2017 Sep;127(3):532-536. doi: 10.3171/2016.8.JNS16538. Epub 2016 Dec 2. PMID 27911234
- [Background] Alan N, Lee P, Ozpinar A, Gross BA, Jankowitz BT. Robotic Stereotactic Assistance (ROSA) Utilization for Minimally Invasive Placement of Intraparenchymal Hematoma and Intraventricular Catheters. World Neurosurg. 2017 Dec;108:996.e7-996.e10. doi: 10.1016/j.wneu.2017.09.027. Epub 2017 Sep 14. PMID 28919568
- [Background] Wang A, Tenner MS, Tobias ME, Mohan A, Kim D, Tandon A. A Novel Approach Using Electromagnetic Neuronavigation and a Flexible Neuroendoscope for Placement of Ommaya Reservoirs. World Neurosurg. 2016 Dec;96:195-201. doi: 10.1016/j.wneu.2016.08.127. Epub 2016 Sep 5. PMID 27609447